CLINICAL TRIAL: NCT00354978
Title: Phase II Study of Irinotecan, Leucovorin, 5-Fluorouracil (FOLFIRI) Plus Bevacizumab as First-Line Treatment for Metastatic Colorectal Cancer
Brief Title: Study of FOLFIRI Plus Bevacizumab in Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0614
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Results first posted 2011-10-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; FOLFIRI; Irinotecan; CPT-11; Leucovorin; LV; Folinic Acid; Fluorouracil; 5-FU; Adrucil; Efudex; Bevacizumab; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI plus Bevacizumab (Experimental): FOLFIRI [folinic acid (leucovorin) 400 mg/m^2 by vein (IV) Day 1; 5-FU 400 mg/m^2 IV injection Day 1 immediately followed by 2.4 g/m^2 IV over 46 hours over Days 1-3; Irinotecan 180 mg/m^2 IV on Day 1] + Bevacizumab 5 mg/kg over 90 minutes on Day 1 administered alone then 5 mg/kg IV on Day 1 of 14 day cycle.
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Leucovorin; Drug: Irinotecan

INTERVENTIONS:
Drug: 5-Fluorouracil — 400 mg/m^2 injection by vein Day 1 of 14 day cycle immediately after completion of leucovorin infusion.
  2.4 g/m^2 by vein over 46 hours over Days 1-3 of 14 day cycle immediately after completion of 400 mg/m^2 injection.
  Other Names: F of FOLFIRI; 5-FU; Adrucil; Efudex
Drug: Bevacizumab — 5 mg/kg over 90 minutes on Day 1 of first 14 day cycle as initial dose, administered alone without other drugs.
  5 mg/kg by vein on Day 1 of 14 day cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Leucovorin — 400 mg/m^2 over 2-4 minutes by vein on Day 1 of 14 day cycle.
  Other Names: FOL of FOLFIRI; LV; folinic acid
Drug: Irinotecan — 180 mg/m^2 by vein over 90 minutes on Day 1 of 14 day cycle.
  Other Names: IRI of FOLFIRI; CPT-11

SUMMARY:
Objectives:

1. To estimate progression-free survival (PFS) at 12 months in subjects with metastatic colorectal cancer who receive FOLFIRI [folinic acid (leucovorin or LV), 5-Fluorouracil (5-FU), irinotecan) plus bevacizumab as first line treatment.
2. To determine the objective response rate and the duration of objective response in this population.
3. To assess overall survival (OS) in this population.
4. To measure the effect of treatment on intratumoral blood volume and microvascular permeability by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) in consenting patients in whom it is technically feasible.
5. To correlate plasma proteomics with response.
6. To assess the safety of this regimen.

DETAILED DESCRIPTION:
Colorectal cancer growth may be affected by a protein in the body called "vascular endothelial growth factor" (VEGF). A drug that blocks VEGF may be an effective treatment for colorectal cancer. Bevacizumab is designed to block VEGF. Bevacizumab will be added to 5-Fluorouracil (5-FU), leucovorin (LV), and irinotecan, a drug combination routinely used in the treatment of advanced colorectal cancer.

Before you can start treatment on the study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will be asked questions about your medical history and about any medications you are currently taking or have taken in the past. You will have a complete physical exam and your heart rate, temperature, breathing rate, blood pressure, height, and weight will be measured. You will be asked about your ability to perform every day activities. You will have an electrocardiogram (ECG - a test that measures the electrical activity of the heart). You will have a chest x-ray and scans (either computed tomography (CT) or magnetic resonance imaging (MRI)) of your abdomen and pelvis to evaluate the cancer. Scans of other parts of your body also may be taken if your doctor thinks they are needed to evaluate your cancer. Blood (about 3 tablespoons) and urine samples will be collected for routine tests, including complete blood count, carcinoembryonic antigen (CEA) level (a marker for your cancer), and chemistry profile. Women who are able to have children must have a negative blood or urine pregnancy test

If the screening evaluations show you are eligible to take part in the study, you may begin treatment Study treatment is repeated every 2 weeks (14 days). Each 14-day period of treatment is called a "cycle" of therapy. You must receive study treatment at M. D. Anderson.

All study drugs will be given through a needle into a vein. For your first treatment, you will receive bevacizumab alone first. The first dose of bevacizumab will be given over about 90 minutes. If you do not have a reaction (such as fever/chills), the next dose will be given over about 60 minutes, and if again no reaction occurs, each dose after that will be given over about 30 minutes. If you experience a reaction to the bevacizumab infusion, you may be given acetaminophen (such as Tylenol) by mouth and/or an antihistamine by vein over 30 minutes before each dose to help decrease the risk of further reactions.

Fourteen (14) days later and for all future cycles, you will receive bevacizumab, LV, and irinotecan given on Day 1 of each cycle. 5-FU is given over 46 hours over Days 1-3.

Bevacizumab will be given as described above. When the bevacizumab infusion ends, you will receive LV and irinotecan, starting at the same time. You will receive irinotecan over 90 minutes and LV over 2 hours. When the LV infusion ends, 5-FU will be given over 2 to 4 minutes. This is followed by more 5-FU given over 46 hours using a small portable pump (about the size of a standard paperback book).

Before each new cycle of study treatment, you will be asked questions about any side effects you may have had and about any medications you are currently taking or have taken since you last saw the study doctor. You will have a complete physical exam, including measurements of blood pressure, pulse, temperature, and weight. You will be asked about your ability to perform every day tasks. About 3 tablespoons of blood will be taken for routine laboratory tests. These tests include a complete blood count and chemistry profile. A urine sample will be taken before every other cycle of treatment. During the first cycle of treatment, on Day 8, you will have a sample of blood (about 3 teaspoons) drawn. This test may be done at a lab close to your home.

You will also have either CT scans or MRI of the tumor(s) every 8 weeks and at the end of the study treatment. About 1 tablespoon of blood will be taken to check your CEA level at the same time scans are done. Additional tests may be done during the study if your doctor feels it is necessary for your care. Except for the weekly blood test, which may be done at a lab close to home, all testing and evaluations must be done at M. D. Anderson.

If you experience severe side effects, treatment may be delayed, stopped, or you may receive smaller doses of the treatment. You may continue to receive study treatment unless the disease gets worse, you decide not to take part any longer, or your doctor decides it is in your best interest to stop treatment.

When you stop study treatment, you will be asked to have some tests and evaluations done at an end of study visit. Urine and about 3 tablespoons of blood will be taken for routine laboratory tests, including complete blood count, CEA level, and chemistry profile. You will also have a physical exam. CT scan or MRI scan of your abdomen and pelvis will also be done to check the size and location of your disease.

Once you stop receiving study treatment, the study doctor or nurse will continue to check how you are doing, either in the clinic or by telephone if you stop coming to M. D. Anderson, every 3 months for the rest of your life.

This is an investigational study. The drugs used in this study are approved by the FDA for treatment of advanced colorectal cancer. Up to 43 patients will take part in this multicenter study. About 38 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically or cytologically confirmed colorectal adenocarcinoma with metastatic disease documented on diagnostic imaging studies.
2. Patient must have measurable lesions as defined by modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Patients who agree to undergo the optional Dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) studies must have a metastatic liver lesion that is > 2 cm.
3. Patient has not previously received chemotherapy for metastatic disease.
4. Patient may have received adjuvant therapy for primary colorectal cancer provided that at least 6 months have elapsed from the time the adjuvant therapy was concluded and recurrent disease was documented.
5. Written informed consent obtained.
6. Age greater than/equal to 18 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
8. Patients must have adequate organ and marrow function as defined below: · Absolute neutrophil count (ANC) greater than/equal to 1,500/mm3; platelets greater than/equal to 100,000/ mm3; hemoglobin greater than/equal to 9 gm/dL (may be transfused to maintain or exceed this level); total bilirubin less than/equal to 1.5 within institutional upper limit of normal (IULN); aspartate aminotransferase (AST or SGOT)/alanine aminotransferase (ALT or SGPT) less than/equal to 2.5 times IULN, or less than/equal to 5 times IULN if known liver metastases; serum creatinine less than/equal to 1.5 times IULN
9. Patients must have an International Normalized Ratio (INR) less than/equal to 1.5 and a Partial thromboplastin time (PTT) less than/equal to IULN
10. Patients with history of hypertension must be well-controlled (blood pressure less than/equal to 150/100), on a stable regimen of anti-hypertensive therapy.

Exclusion Criteria:

1. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental therapeutic drug study other than this protocol.
2. Prior full field radiotherapy less than/equal to 4 weeks or limited field radiotherapy less than/equal to 2 weeks prior to treatment.
3. History or presence of central nervous system metastases.
4. Female patients who are pregnant or lactating or men and women of reproductive potential not willing to employ an effective method of birth control during treatment and for 3 months after discontinuing study treatment.
5. A history of prior treatment with bevacizumab or other agents targeting Vascular endothelial growth factor (VEGF).
6. Known dihydropyrimidine dehydrogenase deficiency.
7. Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, irinotecan, 5-FU, or leucovorin.
8. Serious non-healing wound, ulcer, or active bone fracture.
9. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 0; anticipation of need for major surgical procedure during the course of the study.
10. Fine needle aspirations or core biopsies within 7days prior to Day 0.
11. For patients who agree to Optional DCE-MRI studies: Cardiac pacemaker, neurostimulator, metal implants other than those specifically approved as safe for use in MR scanners at the magnetic field strength used for these studies, claustrophobia, obesity (weight exceeding equipment limits).
12. Current or recent use of full-dose warfarin (except as required to maintain patency of preexisting, permanent indwelling IV catheters) for subjects receiving warfarin, INR should be < 1.5). Patients may have prophylactic use of low molecular weight heparin, however therapeutic use of heparin or low molecular weight heparin is not acceptable.
13. Evidence of bleeding diathesis or coagulopathy.
14. Patients with a history of another primary malignancy less than/equal to 5 years, with the exception of non-melanoma skin cancer, and carcinoma in situ of uterine cervix.
15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0, unless affected area has been removed surgically.
16. Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study: Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen; Unstable angina; New York Heart Association (NYHA) greater than/equal to grade 2 congestive heart failure
17. Myocardial infarction within 6 months of study enrollment; History of stroke within 6 months of study enrollment; Unstable symptomatic arrhythmia requiring medication (Patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible); Clinically significant peripheral vascular disease; Uncontrolled diabetes; Serious active or uncontrolled infection
18. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
19. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 13, 2005 through January 31, 2007. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Forty nine (49) patients were enrolled onto the study, and 6 patients did not meet inclusion criteria and were excluded.
Period: Overall Study
Arm/Group | FOLFIRI Plus Bevacizumab
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FOLFIRI Plus Bevacizumab
Number analyzed (Participants) | 43
Age Continuous [Median (Full Range); unit: years] | 57 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of disease progression using Kaplan-Meier median PFS time.
Time Frame: From baseline until first documented progression or death from any cause, whichever came first, assessed up to 75 months
Population: Analysis per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFIRI Plus Bevacizumab
Number analyzed (Participants) | 43
Months | 12.8 (.02) [9.6 to 15.2]

ADVERSE EVENTS:
Time Frame: 3 years and 4 months
Arm/Group | FOLFIRI Plus Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 43/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI Plus Bevacizumab (N=43)
ALT,SGPT (Serum Glutamic Pyruvic Transaminase) (Metabolism and nutrition disorders) | 9
Abdominal Pain (Gastrointestinal disorders) | 7
Alkaline Phosphatase (Metabolism and nutrition disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 22
Constipation (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 19
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 5
Headache (General disorders) | 10
Hemoglobin (Blood and lymphatic system disorders) | 19
Hemorrhage (Rectum) (Gastrointestinal disorders) | 6
Hemorrhage, Pulmonary (Nose) (Respiratory, thoracic and mediastinal disorders) | 19
Hot Flashes (Reproductive system and breast disorders) | 10
Hypertension (Metabolism and nutrition disorders) | 8
Mucositis (Oral Cavity) (General disorders) | 11
Nausea (Gastrointestinal disorders) | 19
Neuropathy (Sensory) (General disorders) | 7
Neutrophils/Granulocytes (ANC/AGC) (Metabolism and nutrition disorders) | 14
Pain (Muscle) (General disorders) | 12
Proteinuria (Metabolism and nutrition disorders) | 11
Pulmonary (Other) (Respiratory, thoracic and mediastinal disorders) | 5
Serum Glutamic Oxaloacetic Transaminase (AST) (General disorders) | 18
Sweating (General disorders) | 5
Thrombosis (Embolism) (Vascular disorders) | 5
Vomiting (Gastrointestinal disorders) | 16
Watery Eye (Eye disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes